CLINICAL TRIAL: NCT00175643
Title: Open-Label Study to Assess Safety and Efficacy of Imiquimod 5% Cream Applied 3 Days Per Week in 1 or 2 Cycles for Treatment of Actinic Keratoses on the Head
Brief Title: Safety and Efficacy of Imiquimod Applied in Dose-Cycle for Actinic Keratoses
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Vancouver Coastal Health Research Institute (Other); 3M (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK-IMIQUIMOD CYCLING
Record Dates: First submitted 2005-09-11; First posted 2005-09-15 (Estimated); Last update posted 2006-05-09 (Estimated); Status verified 2006-05

CONDITIONS: Actinic Keratoses
Keywords: actinic keratoses; imiquimod; pre-malignant; squamous cell carcinoma; immunosuppression
MeSH Terms: conditions — Keratosis, Actinic; Precancerous Conditions; Carcinoma, Squamous Cell | interventions — Imiquimod

INTERVENTIONS:
Drug: imiquimod

SUMMARY:
It is believed that imiquimod 5% cream has the potential to be an effective treatment for actinic keratoses. The purpose of this study is to evaluate the duration of the effect of topical imiquimod 5% topical cream for the treatment of actinic keratoses.

DETAILED DESCRIPTION:
This study will assess the safety and efficacy of imiquimod 5% cream applied to actinic keratoses on the head to reduce the size of lesions. The objective is to analyze the effect of dose cycling with respect to the complete clearance rate when imiquimod 5% cream is applied 3 times per week for 4 weeks in 1 or 2 cycles. The complete clearance rate is defined as the proportion of subjects with no clinically visible AK lesions in the treatment area at the end of cycle 1 or the end of cycle 2.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* Have a total of 4 to 8 clinically typical, discrete, non-hyperkeratotic, non-hypertrophic AK lesions located within a contiguous 25 cm2 treatment area (balding scalp or face, but not both).
* Free of any significant findings (e.g. tattoos) in the potential application site area that may impair examination of treatment or surrounding area.
* Willing to eliminate tanning bed/sun parlor use for duration of study.

Exclusion Criteria:

* Evidence of clinically significant, unstable cardiovascular or immunosuppressive, hematologic, hepatic, neurologic, renal, endocrine, collagen-vascular, or gastrointestinal abnormalities or disease.
* Any dermatological disease and or condition in the treatment or surrounding area that may be exacerbated by treatment with imiquimod or cause difficulty with examination (e.g. rosacea, psoriasis, atopic dermatitis, eczema).
* Confirmed SCC, BCC anywhere on the head.
* Share a household where there is a person participating in a concurrent clinical study of imiquimod or being treated with imiquimod 5% topical cream.
* Active chemical dependency or alcoholism, as assessed by investigator.
* Females who are pregnant, breast-feeding or considering becoming pregnant while on the study.
* Females with childbearing unwilling to practice an effective method of contraception, as defined by the investigator for the duration of the study as well as one month after completion.
* Received any treatment, products or procedures within the designated time period prior to the prestudy visit as listed on page 4 of the protocol (Version 03 dd March 2003).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2005-02; Study Completion 2005-11

PRIMARY OUTCOMES:
Complete clearance rate - defined as the proportion of subjects at the end of cycle 1 or cycle 2 with no (zero) clinically visible AK lesions in the treatment area.

SECONDARY OUTCOMES:
Partial clearance rate - defined as the proportion of subjects at the end of cycle 2 with at least 75% reduction from the number of AK lesions counted at baseline in the treatment area
Sustained clearance rate at week 8 post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jason K Rivers, M.D., Principal Investigator — Division of Dermatology, University of British Columbia
Locations (1):
- Clinical Trials Unit, Skin Care Centre, UBC Dermatology, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] (1.) Somani N, Rivers JK. Imiquimod 5% cream for the treatment of actinic keratoses. Skin Therapy Lett 2005;10(2):1-6. (2.) Rivers JK. Topical 3% diclofenac in 2.5% hyaluronan gel for the treatment of actinic keratoses. Skin Therapy Lett 2004;9(1):1-3. (3.) Rivers JK, Arlette J, Shear N, Guenther L, Carey W, Poulin Y. Topical treatment of actinic keratoses with 3.0% diclofenac in 2.5% hyaluronan gel. Br J Dermatol 2002;146 (4.) Rivers JK, McLean DI. An open study to assess the efficacy and safety of topical 3% diclofenac in a 2.5% hyaluronic acid gel for the treatment of actinic keratoses. Arch Dermatol 1997;133(10):1239-42.